CLINICAL TRIAL: NCT02717416
Title: Hemostatic Powder Following Injection Therapy Versus Conventional Dual Therapy for Endoscopic Hemostasis for Non-variceal Upper Gastrointestinal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0027
Record Dates: First submitted 2016-03-18; First posted 2016-03-23 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: upper gastrointestinal bleeding; endoscopic hemostasis; hemostatic powder
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Surgical Instruments

STUDY DESIGN:
Intervention Model Description: After randomization, patients in both group will undergo endoscopic hemostasis with epinephrine injection therapy. In the study group, Endo-clot will be applied after epinephrine injection therapy. In the control group, hemoclip will be applied after epinephrine injection therapy. The efficacy of Endo-Clot and hemoclip will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endo-clot™ (EndoClot Plus, Unc., Santa Clara, CA, USA) group (Experimental): The intervention group
  Interventions: Device: Endo-Clot
- Hemoclip (HX-610-135, Olympus, Japan) or electrical coagulation group (Active Comparator): Patients in the control group will undergo endoscopic hemostasis with combination therapy, epinephrine injection therapy and hemoclip or electrical coagulation therapy.
  Interventions: Device: hemoclip or electrical coagulation

INTERVENTIONS:
Device: Endo-Clot — After epinephine injection therapy, Endo-Clot is applied immediately onto the bleeding lesion. A total of 2 g of AMP® particle powder will be sprayed onto the bleeding lesion by a catheter inserted through a working channel of the endoscope under continuous air flow.
  Other Names: Hemostatic powder group
  Arms: Endo-clot™ (EndoClot Plus, Unc., Santa Clara, CA, USA) group
Device: hemoclip or electrical coagulation — After epinephrine injection therapy, hemoclip (HX-610-135, Olympus, Japan) will be applied onto the bleeding lesions. The number of hemoclip will be decided by endoscopist. Electrical coagulation will be applied onto the bleeding lesions.
  Other Names: Mechanical therapy (clip) or electrical coagulation group
  Arms: Hemoclip (HX-610-135, Olympus, Japan) or electrical coagulation group

SUMMARY:
Acute upper gastrointestinal hemorrhage (UGIH) is a common condition that leads to hospital admission, and has significant associated morbidity and mortality, especially in the elderly. The most common causes of acute UGIH are nonvariceal. Although up 70% of non-variceal bleeds settle with conservative measures, endoscopic therapy is the established method for treating those bleeds for which this is not sufficient. Despite advances and increased expertise in managing upper gastrointestinal bleeding, the associated mortality of up to 15% has remained unchanged for several years.

EndoClot is a novel topical hemostatic powder approved for use in non-variceal upper gastrointestinal bleeding. This study examines its efficacy for endoscopic hemostasis in non-variceal upper gastrointestinal bleeding. This is a multicenter, prospective, randomized study.

DETAILED DESCRIPTION:
Patients with upper GI bleeding who need endoscopic hemostasis will be enrolled in this study. When there is a upper GI bleeding with active bleeding or stigmata on the lesions, endoscopic hemostasis will be done.

After randomization, patients in both group will undergo endoscopic hemostasis with epinephrine injection therapy. In the study group, Endo-clot will be applied after epinephrine injection therapy. In the control group, hemoclip will be applied after epinephrine injection therapy. The efficacy of Endo-Clot and hemoclip will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 19 years old
2. Patients with hematemesis, hematochezia, melena, suspected upper gastrointestinal bleeding
3. Inpatients who were consulted gastroenterologist for management of upper gastrointestinal bleeding
4. Patients who are planned to undergo EGD for management of upper gastrointestinal bleeding

Exclusion Criteria:

1. Patients who had diagnosed esophageal cancer or stomach cancer
2. Patients who are suspected variceal bleeding, had medical history of liver cirrhosis, hepatocellular carcinoma
3. Coagulation disorder (hemophilia, ITP,,)
4. Post-procedure bleeding (EGD biopsy, EMR, ESD, stent insertion..)
5. Patients who cannot undergo EGD because of anatomical problem, unconsciousness.
6. Patients who are unwilling or unable to provide informed consent, such as those with psychiatric problem, drug abuse or alcoholism

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
The rate of successful initial hemostasis | 5 minites after appilication of Endo-Clot
  The primary endpoint was immediate hemostasis which defined as endoscopic observation of bleeding cessation for 5 minutes after appilication of Endo-Clot.

SECONDARY OUTCOMES:
Rebleeding rates | 0~14 days after initial endoscopic hemostasis
  The secondary endpoint was rebleeding rates within 14 days. Rebleeding is defineds as clinical presentation of hematemesis, melena or hematochezia.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university of medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share data

REFERENCES:
- [Derived] Jung DH, Park CH, Choi SI, Kim HR, Lee M, Moon HS, Park JC. Comparison of a Polysaccharide Hemostatic Powder and Conventional Therapy for Peptic Ulcer Bleeding. Clin Gastroenterol Hepatol. 2023 Oct;21(11):2844-2853.e5. doi: 10.1016/j.cgh.2023.02.031. Epub 2023 Mar 10. PMID 36906081